CLINICAL TRIAL: NCT05229497
Title: A Phase Ib/II Study of AK112#PD-1/VEGF Bispecific Antibody# in Combination With AK117#Anti-CD47 Antibody# in Advanced Malignant Tumors
Brief Title: A Phase Ib/II Study of AK112 in Combination With AK117 in Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK117-201
Record Dates: First submitted 2022-01-28; First posted 2022-02-08 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Advanced Malignant Tumors
MeSH Terms: interventions — Carboplatin; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase Ib#Dosage regimen 1# (Experimental): Subjects receive AK112 (20 mg/kg Q3W) + AK117 (30 mg/kg QW)
  Interventions: Drug: AK112; Drug: AK117
- Phase Ib#Dosage regimen 2# (Experimental): Subjects receive AK112 (20 mg/kg Q3W) + AK117 (45 mg/kg QW)
  Interventions: Drug: AK112; Drug: AK117
- Phase II#Cohort 1# (Experimental): Head and neck squamous cell carcinoma (HNSCC): AK112 (20 mg/kg Q3W)
  Interventions: Drug: AK112
- Phase II#Cohort 2# (Experimental): HNSCC: AK112 (20 mg/kg Q3W) + AK117 (recommended Phase 2 dose)
  Interventions: Drug: AK112; Drug: AK117
- Phase II#Cohort 3# (Experimental): HNSCC: AK112 (20 mg/kg Q3W) + AK117 (recommended Phase 2 dose)+Carboplatin/cisplatin+5-fluorouracil
  Interventions: Drug: AK112; Drug: AK117; Drug: Carboplatin; Drug: Cisplatin; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: AK112 — IV infusion,Specified dose on specified days
Drug: AK117 — IV infusion,Specified dose on specified days
  Arms: Phase II#Cohort 2#; Phase II#Cohort 3#; Phase Ib#Dosage regimen 1#; Phase Ib#Dosage regimen 2#
Drug: Carboplatin — IV infusion,Specified dose on specified days
  Arms: Phase II#Cohort 3#
Drug: Cisplatin — IV infusion,Specified dose on specified days
  Arms: Phase II#Cohort 3#
Drug: 5-Fluorouracil — IV infusion,Specified dose on specified days
  Arms: Phase II#Cohort 3#

SUMMARY:
Phase Ib/II open label, multicenter study to evaluate the efficacy and safety of AK112 (anti-PD-1 and VEGF bispecific antibody) combined with AK117#AntiCD47 Antibody# in advanced malignant tumors

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years old.
2. Have a life expectancy of at least 3 months.
3. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Phase Ib: Histologically or cytologically confirmed selected advanced solid tumor.
5. Phase II:

   Cohort 1 and 2 :

   A. Has histologically confirmed recurrent or metastatic HNSCC who had failed only first-line platinum-containing therapy.

   B. Has histologically confirmed recurrent or metastatic HNSCC with PD-L1 positive (CPS≥1) without prior systemic antitumor therapy.

   Cohort 3: Has histologically confirmed recurrent or metastatic HNSCC without prior systemic antitumor therapy.
6. Have at least one measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by investigator.
7. Has adequate organ function.

Exclusion Criteria:

1. Undergone major surgery within 30 days prior to the first dose of study treatment.
2. Active central nervous system (CNS) metastases.
3. History of active autoimmune disease that has required systemic treatment in the past 2 years (i.e.,corticosteroids or immunosuppressive drugs).
4. Active Hepatitis B or Hepatitis C.
5. Received previous immunotherapy, including immune checkpoint inhibitors, immune checkpoint agonists, immune cell therapy and other treatments targeting the mechanism of tumor immunity.
6. History of severe bleeding tendency or coagulation disorder.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Adverse Events (AEs) | Up to approximately 2 years
  Characterization of incidence, severity and abnormal clinically significant laboratory findings of AEs
Number of patients experiencing dose-limiting toxicities (DLTs) | During the first 3 weeks
Objective Response Rate (ORR) | Up to approximately 2 years

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to approximately 2 years
Duration of Response (DOR) | Up to approximately 2 years
Time to response (TTR) | Up to approximately 2 years
Progression free survival (PFS) | Up to approximately 2 years
Overall survival (OS) | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Chen, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China